CLINICAL TRIAL: NCT02848378
Title: The Levels of Advanced Oxidation Protein Product and Monocyte Chemoattractant Protein-1 in Gingival Crevicular Fluid in Periodontal Disease and Health
Brief Title: Advanced Oxidation Protein Product and Monocyte Chemoattractant Protein-1 in Periodontal Disease
Status: Completed | Type: Observational
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Meltem Karsiyaka Hendek, Corresponding author, Clinical Research, Kırıkkale University
Other Study IDs: 2014/17
Record Dates: First submitted 2016-07-21; First posted 2016-07-28 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Inflammation; Periodontal Disease
Keywords: Advanced Oxidation Protein Products; Gingival crevicular fluid; Monocyte chemoattractant protein-1; Periodontal Disease
MeSH Terms: conditions — Inflammation; Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Chronic periodontitis group: Subjects who have moderate to severe alveolar bone loss and clinical attachment level (CAL) ≥5 mm and probing depth (PD) ≥6mm in multiple sites of all four quadrants of the mouth but with no evidence of rapid progression
- Gingivitis group: Subjects who show gingival inflammation that is based on the presence of bleeding on probing (BOP) at >50% of sites in the whole mouth, no clinical and radiographic signs of periodontitis
- Periodontally healthy group: Subjects who have no sites with PD >3mm and CAL >0 mm, a BOP score of <15% at the examination and no alveolar bone loss.

SUMMARY:
This study investigates the levels of advanced oxidation protein product and monocyte chemoattractant protein-1 in gingival crevicular fluid in periodontal disease and health. 25 participants with chronic periodontitis, 25 participants with gingivitis and 25 periodontally healthy subjects are included into this study. In each participant, four sites are identified for gingival crevicular fluid samples.

DETAILED DESCRIPTION:
Oxidative stress is the disequilibrium between the formation of free radicals and antioxidant defense mechanisms via damaging cellular macromolecules (DNA, protein, lipid, etc..) which are susceptible to oxidative damage.

Advanced oxidation protein product is identified as a new marker of protein oxidation.

Monocyte chemoattractant protein-1 is a major chemoattractant for lymphocytes, monocytes and macrophages.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic periodontitis and gingivitis

Exclusion Criteria:

* Systemic illnesses
* Any medications known to affect the periodontium
* Pregnancy and lactation

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 25 participants with chronic periodontitis, 25 participants with gingivitis and 25 periodontally healthy subjects are included.
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2014-05; Primary Completion 2015-01 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Advanced oxidation protein product (nmol) | Before periodontal treatment

SECONDARY OUTCOMES:
Monocyte chemoattractant protein-1(pg) | Before periodontal treatment
The probing depth (mm), clinical attachment level (mm), plaque index scores (0-3) and gingival index scores (0-3) | Before periodontal treatment

IPD SHARING:
Plan to Share IPD: No